CLINICAL TRIAL: NCT04620135
Title: A Single-masked, Randomized, Multi-center, Parallel-group, 4-week Study Evaluating the Efficacy and Safety of Once Daily Netarsudil Ophthalmic Solution 0.02% Compared to Twice Daily Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4% in Japanese Subjects With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Brief Title: Efficacy and Safety Study of Netarsudil 0.02% Ophthalmic Solution Compared to Ripasudil Hydrochloride Hydrate 0.4% Ophthalmic Solution in Japanese Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-13324-CS305
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma, Primary Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study adopted a single-masked study design. Treatment assignments were masked to the Investigator, the clinical study team (Sponsor, designated personnel involved in day-to-day study management, Monitors, Data Managers, and Statisticians), and the subjects for the duration of the study. The netarsudil and ripasudil bottles were different in the study, however, investigators and subjects were masked to study drug assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netarsudil ophthalmic solution 0.02% and netarsudil ophthalmic solution vehicle (Experimental): 1 drop netarsudil 0.02% in the evening and 1 drop netarsudil vehicle in the morning in each eye.
  Interventions: Drug: Netarsudil ophthalmic solution 0.02%
- Ripasudil hydrochloride hydrate ophthalmic solution 0.4% (Active Comparator): 1 drop ripasudil twice daily in the morning and evening in each eye.
  Interventions: Drug: Ripasudil hydrochloride hydrate ophthalmic solution 0.4%

INTERVENTIONS:
Drug: Netarsudil ophthalmic solution 0.02% — Topical sterile ophthalmic solution Other Name: Rhopressa®
  Other Names: Vehicle: Netarsudil ophthalmic solution
  Arms: Netarsudil ophthalmic solution 0.02% and netarsudil ophthalmic solution vehicle
Drug: Ripasudil hydrochloride hydrate ophthalmic solution 0.4% — Other Name: Glanatec®
  Arms: Ripasudil hydrochloride hydrate ophthalmic solution 0.4%

SUMMARY:
A Phase 3 Study Comparing the Efficacy and Safety of Netarsudil Ophthalmic Solution 0.02% QD to Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4% BID, for Treatment of Primary Open-Angle Glaucoma or Ocular Hypertension Over A 4-Week Period.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Diagnosis of POAG or OHT in both eyes (POAG in one eye and OHT in the fellow eye was acceptable)
* Medicated intraocular pressure (IOP) ≥ 14 mmHg in at least one eye and < 30 mmHg in both eyes at screening visit
* For POAG eyes, unmedicated (post washout) IOP ≥ 15 mmHg and < 35 mmHg in the study eye at 2 qualification visits (09:00 hours), 2-7 days apart. At second qualification visit IOP ≥ 15 mmHg and < 35 mmHg at 11:00 and 16:00 hour (in the same eye).
* For OHT eyes, unmedicated (post washout) IOP ≥ 22 mmHg and < 35 mmHg in the study eye at 2 qualification visits (09:00 hours), 2-7 days apart. At second qualification visit IOP ≥ 22 mmHg and < 35 mmHg at 11:00 and 16:00 hours (in the same eye)
* Best-corrected visual acuity (BCVA) +0.7 log MAR or better (20/100 Snellen or better or 0.20 or better in decimal unit) in each eye
* Willingness and ability to give signed informed consent and follow study instructions

Exclusion Criteria:

* Clinically significant ocular disease
* Retinal diseases that may progress during the study period
* Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure glaucoma, or narrow angles
* Previous glaucoma intraocular surgery
* Refractive surgery in either eye
* Ocular hyperemia score of moderate (+2) or severe (+3) at Qualification Visit #2
* Ocular trauma
* Ocular infection or inflammation
* Any corneal disease that may confound assessment
* Evidence of corneal deposits or cornea verticillata
* Known hypersensitivity to any component of netarsudil ophthalmic solution 0.02%, ripasudil hydrochloride hydrate ophthalmic solution 0.4%, or to topical anesthetic.
* Mean central corneal thickness >620 um
* Any abnormality preventing reliable Goldmann applanation tonometry of either eye (e.g. keratoconus)
* Cannot demonstrate proper delivery of the eye drop
* Clinically significant systemic disease
* Participation in any investigational study within 30 days prior to screening
* Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joella Kittrell, Study Director — Aerie Pharmaceuticals
Locations (1):
- Seijo Clinic, Setagaya-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Araie M, Sugiyama K, Aso K, Kanemoto K, Iwata R, Hollander DA, Senchyna M, Kopczynski CC. Phase 3 Clinical Trial Comparing the Safety and Efficacy of Netarsudil to Ripasudil in Patients with Primary Open-Angle Glaucoma or Ocular Hypertension: Japan Rho Kinase Elevated Intraocular Pressure Treatment Trial (J-ROCKET). Adv Ther. 2023 Oct;40(10):4639-4656. doi: 10.1007/s12325-023-02550-w. Epub 2023 Aug 21. PMID 37603205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at 27 clinic sites in Japan starting on 30Nov2020 with last subject last visit on 30July2021.
Pre-assignment Details: Subjects were required to washout of their pre-study ocular hypotensive medication for a prescribed period as specified in the protocol prior to attending Qualification Visit #1.
Period: Intent-to-Treat (ITT) Population
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Started | 122 | 123
Completed | 118 | 120
Not Completed | 4 | 3
Period: Per-Protocol (PP) Population
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Started | 121 | 122
Completed | 117 | 119
Not Completed | 4 | 3
Period: Safety Population
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Started | 122 | 123
Completed | 118 | 120
Not Completed | 4 | 3
Period: Study Completion
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Started | 122 | 123
Completed | 118 | 120
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4% | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 65 years | 63 | 60 | 123
  Age Category: >= 65 years | 59 | 63 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 66 | 144
  Male | 44 | 57 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Study Eye Diagnosis [Count of Participants; unit: Participants]
  Ocular Hypertension | 32 | 35 | 67
  Primary Open Angle Glaucoma | 90 | 88 | 178

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Comparison of both groups mean diurnal IOP at Week 4 (Day 29). IOP will be measured by Goldmann applanation tonometry and reported in millimeters mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Mean diurnal IOP was calculated as the average of 3 IOP values across 09:00, 11:00 and 16:00 time points.
Time Frame: 29 Days
Population: The intent-to-treat (ITT) population was used for the primary analysis of the efficacy variables and included all randomized subjects (as randomized) who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Number analyzed (Participants) | 122 | 123
mmHg | 15.96 (0.157) | 17.71 (0.155)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle vs Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%; Test type: Superiority; p < 0.00001, ANCOVA — Analyzed as ANCOVA with mean diurnal IOP at Week 4 as the response, baseline mean diurnal IOP as a covariate, and treatment as a main effect, using the ITT population with MCMC and regression-based multiple imputation to impute missing data; The least squares (LS) mean difference = -1.74, 95% CI 2-sided [-2.17 to -1.31], Standard Error of Mean 0.221; The primary analysis of the primary endpoint employed an analysis of covariance (ANCOVA) with mean diurnal IOP at Week 4 as the response, baseline mean diurnal IOP as a covariate, and treatment as a main effect, using the ITT population with Markov Chain Monte Carlo (MCMC) and regression based multiple imputation (MI) techniques to impute missing data. The least squares (LS) mean difference (netarsudil - ripasudil) was presented with a 2-sided p-value and 95% confidence intervals (CIs). A success criterion for the superiority of netarsudil to ripasudil was defined as the 2-sided p value ≤ 0.05 for testing the difference (netarsudil QD - ripasudil BID) to 0 and the point estimate of the LS mean difference of < 0

2. Secondary Outcome: IOP at Weeks 1 and 2
Description: Mean diurnal IOP as measured in mmHg at each post-treatment visit.
Time Frame: Day 8, Day 15
Population: ITT
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Number analyzed (Participants) | 122 | 123
mmHg
  Mean diurnal IOP at Weeks 1 (Days 8) | 16.28 (0.143) | 17.87 (0.141)
  Mean diurnal IOP at Weeks 2 (Days 15) | 16.02 (0.168) | 17.83 (0.166)

3. Secondary Outcome: Mean Change IOP From Baseline at Days 8, 15, 29
Description: Mean change from baseline in mean diurnal IOP as measured in mmHg at each post-treatment visit.
Time Frame: Baseline (Day 1), Days 8, 15, 29
Population: ITT
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
Number analyzed (Participants) | 122 | 123
mmHg
  Baseline IOP mean diurnal IOP | 20.475 (0.2510) | 20.830 (0.3198)
  V4: Week 1 (Day 8) Change from Baseline | -4.341 (0.1603) | -2.814 (0.1397)
  V5: Week 2 (Day 15) Change from Baseline | -4.601 (0.1728) | -2.852 (0.1759)
  V6: Week 4 (Day 29) Change from Baseline | -4.653 (0.1701) | -2.983 (0.1622)

ADVERSE EVENTS:
Time Frame: Volunteered or solicited AEs were collected from the time the subject received the first dose of study medication until Week 4 (Day 29) or study discontinuation. Unresolved AEs at the time of study exit were followed with proper medical care until the event was considered resolved or stabilized, the subject was lost to follow-up, or another resolution to the event was identified.
Description: An overall summary was presented including the number of treatment emergent AEs (TEAEs) and the number and percentage of subjects who experienced at least one TEAE, as well as categorized overall summaries for TEAEs (ocular and non-ocular), TE-SAEs, treatment-related TEAEs and TE-SAEs, TEAEs by maximum severity and by relationship to study drug, TEAEs leading to treatment or study discontinuation, and TEAEs resulting in death.
Arm/Group | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4%
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/122 | 2/123
Other Adverse Events (participants affected / at risk) | 73/122 | 82/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle (N=122) | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4% (N=123)
Infections and infestations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pneumonia
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Erythema multiforme
Treatment-Emergent Serious Adverse Event (TE-SAE) (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Netarsudil Ophthalmic Solution 0.02% and Netarsudil Ophthalmic Solution Vehicle (N=122) | Ripasudil Hydrochloride Hydrate Ophthalmic Solution 0.4% (N=123)
Conjunctival hyperaemia (Eye disorders) | 67 | 77
Eye irritation (Eye disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT04620135/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT04620135/SAP_003.pdf